CLINICAL TRIAL: NCT06806722
Title: Evaluation of Cardiac Mechanics by Speckle Tracking as a Prognostic Tool in Patients With Chagas Cardiomyopathy
Brief Title: Cardiac Mechanics by Speckle Tracking as a Prognostic Predictor in Patients With Chagas Cardiomyopathy
Acronym: ST-Chagas
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto de Cardiologia do Distrito Federal (Other)
Responsible Party: Principal Investigator, Luiz Carlos Madruga Ribeiro, Cardiologist, Echocardiography Specialist, Institute of Cardiology of the Federal District., University of Sao Paulo
Other Study IDs: 40088920.9.3001.0068; 40088920.9.0000.0026 (Other: CAAE)
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chagas Cardiomyopathy; Speckle Tracking Echocardiography; Arrythmias; Sudden Death; ICD
Keywords: Chagas Cardiomyopathy; Speckle Tracking; Global Longitudinal Strain; Mechanical Dispersion; Echocardiography; Heart Failure; Prognostic Markers; Chagas Disease
MeSH Terms: conditions — Chagas Cardiomyopathy; Death, Sudden; Heart Failure; Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1 - Cross Sectional: Patients with an implantable cardioverter defibrillator (ICD) for secondary prevention.
- Group 2 - Cross Sectional: atients without an ICD and no history of severe arrhythmic events. The purpose of this arm is to compare echocardiographic parameters, such as global longitudinal strain (GLS) and mechanical dispersion (MD), between high-risk and lower-risk patients.
- Longitudinal Cohort: This cohort includes all patients from the cross-sectional phase, who will be prospectively followed for 24 months to evaluate clinical outcomes.

SUMMARY:
This study aims to evaluate the prognostic value of myocardial mechanics parameters, including global longitudinal strain (GLS) and mechanical dispersion (MD), assessed through speckle tracking echocardiography, in patients with Chagas cardiomyopathy (CCM). The study is divided into two arms: a cross-sectional arm and a longitudinal arm. The cross-sectional arm compares echocardiographic parameters between patients with and without implantable cardioverter defibrillators (ICD) for secondary prevention. The longitudinal arm assesses clinical outcomes over 24 months. Primary outcomes include all-cause mortality and hospitalization due to heart failure, while secondary outcomes encompass sudden cardiac death, sustained ventricular tachycardia, embolic events, and persistent atrial fibrillation.

DETAILED DESCRIPTION:
The study is divided into two phases:

Cross-sectional phase: Patients with CCM and LV ejection fraction (LVEF) ≤50% will be categorized into two groups based on the presence or absence of an ICD for secondary prevention. GLS and MD parameters will be evaluated to determine their association with higher-risk patients.

Longitudinal phase: Patients from the cross-sectional phase will be followed for 24 months to assess primary outcomes (all-cause mortality and heart failure hospitalization) and secondary outcomes (sudden cardiac death, sustained ventricular tachycardia, embolic events, and persistent atrial fibrillation). Prognostic utility of GLS and MD will be compared with traditional parameters.

Study Design:

Study Type: Observational

Estimated Enrollment: 153 participants

Observational Model: Cohort

Time Perspective: Prospective

Study Start Date: [To be added]

Primary Completion Date: [To be added]

Study Completion Date: [To be added]

Outcome Measures:

Primary Outcome Measures:

All-cause mortality (Time Frame: 24 months)

Hospitalization due to heart failure (Time Frame: 24 months)

Secondary Outcome Measures:

Sudden cardiac death (Time Frame: 24 months)

Sustained ventricular tachycardia (Time Frame: 24 months)

Embolic events (Time Frame: 24 months)

Persistent atrial fibrillation (Time Frame: 24 months)

Eligibility Criteria:

Inclusion Criteria:

Age 18-70 years

Diagnosed Chagas disease confirmed by two serological tests

LVEF ≤50% (Simpson's method)

Clinically stable for at least three months

Sinus rhythm or paced atrial rhythm on ECG

Signed informed consent

Exclusion Criteria:

Significant coronary artery disease

End-stage heart failure (Stage D)

Ischemic cardiomyopathy

Severe systemic hypertension

Primary moderate or severe valvular lesions

Inadequate echocardiographic window

Persistent atrial fibrillation or flutter

BMI <18 kg/m² or alcohol consumption >80 g/day

Life expectancy <1 year due to other conditions

Study Arms:

Cross-sectional Group:

Group 1: CCM patients with ICD (high-risk group)

Group 2: CCM patients without ICD

Longitudinal Group:

All patients followed for outcomes.

Statistical Analysis:

Normality of quantitative variables will be tested using the Kolmogorov-Smirnov test.

Differences between groups analyzed using t-tests, Mann-Whitney tests, chi-square tests, or Fisher's exact tests.

Multivariable Cox proportional hazards models will assess predictors of high-risk outcomes.

Kaplan-Meier survival analysis will estimate event-free survival rates.

Sponsor and Collaborators:

Sponsor: Institute of Cardiology, Federal District, Brazil

Collaborators:

Heart Institute (InCor) - University of São Paulo

Santa Lúcia South Hospital

Principal Investigators:

Dr. Luiz Carlos Madruga Ribeiro

Dr. Ludhmila Abrahão Hajjar

Dr. Adenalva Lima de Souza Beck

Funding Source:

Self-funded (Estimated total cost: BRL 8,200)

Ethical Considerations:

Approved by the ethics committee of ICDF.

Confidentiality and participant safety are prioritized.

Echocardiograms performed by trained physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosed Chagas disease confirmed by two serological tests
* LVEF ≤50% (Simpson's method)
* Clinically stable for at least three months
* Sinus rhythm or paced atrial rhythm on ECG
* Signed informed consent

Exclusion Criteria:

* Significant coronary artery disease
* End-stage heart failure (Stage D)
* Ischemic cardiomyopathy
* Severe systemic hypertension
* Primary moderate or severe valvular lesions
* Inadequate echocardiographic window
* Persistent atrial fibrillation or flutter
* BMI <18 kg/m² or alcohol consumption >80 g/day
* Life expectancy <1 year due to other conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with confirmed Chagas cardiomyopathy (CCM) and reduced left ventricular ejection fraction (≤50%) who are clinically stable and receiving outpatient care. Participants will be recruited consecutively from cardiology clinics in the Federal District and surrounding areas. Eligibility criteria ensure a focus on individuals at higher risk of adverse cardiovascular events, while exclusions aim to eliminate confounding factors such as severe comorbidities or inadequate imaging quality. The population represents a cohort of adults aged 18-70 years with confirmed Chagas disease, reflecting the demographic most affected by this condition.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality and Heart Failure Hospitalization | 24 months from the date of enrollment
  The primary outcome measure is a composite endpoint of all-cause mortality and hospitalization due to heart failure over a 24-month follow-up period. Mortality will include any death, regardless of cause. Hospitalization due to heart failure will be defined as an unplanned admission with a primary diagnosis of heart failure requiring intravenous diuretics, inotropic support, or other specialized management for decompensation. These events will be assessed using medical records, patient reports, or direct contact with healthcare providers.

SECONDARY OUTCOMES:
Sudden Cardiac Death | 24 months from the date of enrollment.
  Sudden cardiac death will be defined as death occurring within one hour of symptom onset or when the individual was last seen in stable health within 24 hours prior to death. Events will be confirmed through medical records, autopsy reports, or witness statements.
Sustained Ventricular Tachycardia | 24 months from the date of enrollment.
  ustained ventricular tachycardia will be defined as a ventricular rhythm lasting 30 seconds or more, or requiring termination due to hemodynamic instability. Episodes will be confirmed using ICD/device reports or electrocardiographic documentation.
Embolic Events | 24 months from the date of enrollment.
  Embolic events will include confirmed cases of stroke, transient ischemic attack, or systemic embolism as documented by imaging studies or clinical reports.
Persistent Atrial Fibrillation | 24 months from the date of enrollment.
  Persistent atrial fibrillation will be defined as continuous atrial fibrillation lasting more than 7 days or requiring medical or electrical cardioversion. Diagnoses will be confirmed through electrocardiographic or device reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do DF, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly to ensure participant confidentiality and privacy Data will be analyzed and reported in aggregate form only, in accordance with ethical guidelines and participant consent.

REFERENCES:
- [Background] Carluccio E, Biagioli P, Lauciello R, Zuchi C, Mengoni A, Bardelli G, Alunni G, Gronda EG, Ambrosio G. Superior Prognostic Value of Right Ventricular Free Wall Compared to Global Longitudinal Strain in Patients With Heart Failure. J Am Soc Echocardiogr. 2019 Jul;32(7):836-844.e1. doi: 10.1016/j.echo.2019.02.011. Epub 2019 Apr 9. PMID 30979539
- [Background] Azevedo ACA, Barros MVL, Klaboe LG, Edvardsen T, Costa HS, Paixao GMM, Junior ORS, Nunes MCP, Rocha MOC. Association between myocardial mechanical dispersion and ventricular arrhythmogenicity in chagas cardiomyopathy. Int J Cardiovasc Imaging. 2021 Sep;37(9):2727-2734. doi: 10.1007/s10554-021-02246-8. Epub 2021 Apr 21. PMID 33881664